CLINICAL TRIAL: NCT01284179
Title: Home Hypnotherapy for Refractory Functional Chest Pain: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ryan Madanick, MD, Assistant Professor of Medicine Director, UNC Gastroenterology & Hepatology Fellowship Program, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-0772; R24DK067674 (NIH)
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Functional Chest Pain
Keywords: Functional Chest Pain; Functional GI Disorders; Home Hypnotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypnotherapy (Experimental): Participants will be randomized to either the home hypnotherapy or educational group. The HHT protocol will consist of sequences of two different types of sessions, longer biweekly sessions (LS), each approximately 30-40 minutes in length, and shorter daily sessions (SS), approximately 12 minutes in length. On the first day of each sequence, the patient will listen to the appropriate LS. The patients will listen to the SS on a daily basis in between each LS. Every 2 weeks a new sequence will begin, for a total of 12 weeks of treatment.
  Interventions: Behavioral: Home Hypnotherapy
- Educational (Other): Participants will be randomized to receive either home hypnotherapy or an educational program. The control group will receive an educational digital audio program on MP3 players. These digital audio files will contain general information about FCP and FGIDs. These audio files will be similar to the intervention audio files in length. Patients will be instructed to begin listening on the day of randomization. Patients will be instructed to continue their other medical treatment for chest pain during the study. The control group will be assessed at the same times as the HHT group.
  Interventions: Behavioral: Educational

INTERVENTIONS:
Behavioral: Home Hypnotherapy — Each session contains the following elements: (1) trance induction consisting of narrowing the focus of attention and eye-closure, (2) trance deepening through imagery, guided dissociation from the here-and-now and graded suggestions of change in mental state, (3) vivid guided imagery that engages all the senses and implies improved health, well-being and a sense of strength and personal power, (4) therapeutic suggestions and imagery, both direct and indirect, for enhanced chest comfort, overall physical comfort and mental well-being and immunity to discomfort, that is suggested will last beyond termination of the session and become more noticeable and permanent over time, and (5) trance termination through direct suggestions and counting.
  Arms: Hypnotherapy
Behavioral: Educational — Educational recordings regarding FCP and FGIDs.
  Arms: Educational

SUMMARY:
The primary aim is to develop and test the feasibility of a standardized digital audio home-hypnotherapy (HHT) program for patients with refractory functional chest pain (FCP).

The secondary aims of this study are:

1. To obtain pilot data to assess the magnitude of the treatment effect of self-hypnosis in refractory FCP for an anticipated future, larger treatment trial;
2. To determine the stability of the treatment effect of HHT in refractory FCP;
3. To assess the relationship between response to HHT and psychological factors; and
4. To assess the relationship between response to HHT and symptomatic dimensions of chest pain (severity, frequency, and duration).
5. To assess the difference

DETAILED DESCRIPTION:
Eligible patients with refractory FCP will be randomized to one of 2 arms: the active treatment group, who will receive the HHT program; or a control group. Patients in the active treatment group will receive the 12-week digital audio HHT program. This protocol consists of 7 sessions, each approximately 30-40 minutes, administered every 2 weeks, for a cumulative 12 weeks of treatment, along with a shorter (approximately 12 minute) session administered daily. Patients in the control group will receive a digital audio educational program. Subjects in both groups will be assessed at baseline, 4-6 weeks into treatment, at the end of the treatment, and 3 months after conclusion of the program. Global change in symptoms will be assessed with a 7-point Likert scale. Patients will be considered to respond if they have significant improvement on the Likert scale at the post-treatment visit. Patients will complete a chest pain symptom diary, the SCL-90 and the Coping Strategies Questionnaire-Catastrophizing subscale to assess psychological features, and the SF-36 as a measure of Health Related Quality of Life (HRQOL).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80, male or female.
* Patients must fulfill the Rome III criteria for Functional Chest Pain of Presumed Esophageal Origin for the previous 3 months (with symptom onset at least 6 months before diagnosis), including all of the following:

  * Midline chest pain or discomfort that is not of burning quality
  * Absence of evidence that gastroesophageal reflux is the cause of the symptom
  * Absence of histopathology-based esophageal motility disorders
* Persistent symptoms despite a trial of antidepressant therapy, as defined by either:

  * chest pain despite at least a continuous 4-week trial of at least one antidepressant within the last 6 months; or
  * intolerance of at least one antidepressant within the last 6 months.
* Negative cardiac evaluation (negative cardiac stress test or negative coronary angiogram)
* Negative gastrointestinal evaluation for cause of the pain, defined by absence of Los Angeles grade C or D erosive esophagitis on endoscopy, persistent chest pain on PPI therapy, and no association of chest pain with reflux episodes on an ambulatory pH or pH-impedance study, defined as a symptom index <50% or symptom association probability <95% for chest pain .

Exclusion Criteria:

* Severe co-morbid illness (cardiac, pulmonary, renal, hematologic, hepatic)
* Prior treatment with hypnosis/hypnotherapy for a medical condition
* Prior major thoracic surgery
* Prior diagnosis of or treatment for dissociative disorders, post-traumatic stress disorder, borderline personality disorder, or other psychiatric disorders that include psychotic features
* Pregnancy or planned pregnancy within the upcoming 3 months
* Inability or unwillingness to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Global change in chest pain at the 12 weeks | 12 Weeks Post Treatment Start
  To fulfill Rome III recommendations for the design of treatment trials for Functional Gastrointestinal Disorders (FGIDS),47 we will use a 7-point Likert scale to assess for global change in chest pain. At times V2, V3, and V4, patients will be asked the following question: "Compared to before starting this therapy, how would you rate your chest pain?" The following answers will be given as options: "much better" (+3), "somewhat better" (+2), "minimally better" (+1), "no change" (0), "minimally worse" (-1), "somewhat worse" (-2), "much worse" (-3).

SECONDARY OUTCOMES:
Global change in chest pain at 4 weeks | 4 Weeks Post Treatment Start
  To fulfill Rome III recommendations for the design of treatment trials for Functional Gastrointestinal Disorders (FGIDS),47 we will use a 7-point Likert scale to assess for global change in chest pain. At times V2, V3, and V4, patients will be asked the following question: "Compared to before starting this therapy, how would you rate your chest pain?" The following answers will be given as options: "much better" (+3), "somewhat better" (+2), "minimally better" (+1), "no change" (0), "minimally worse" (-1), "somewhat worse" (-2), "much worse" (-3).
Global change in chest pain at 6 weeks | 6 Weeks Post Treatment Start
  To fulfill Rome III recommendations for the design of treatment trials for Functional Gastrointestinal Disorders (FGIDS),47 we will use a 7-point Likert scale to assess for global change in chest pain. At times V2, V3, and V4, patients will be asked the following question: "Compared to before starting this therapy, how would you rate your chest pain?" The following answers will be given as options: "much better" (+3), "somewhat better" (+2), "minimally better" (+1), "no change" (0), "minimally worse" (-1), "somewhat worse" (-2), "much worse" (-3).
Change in symptom score at 3 months | 12 Weeks Post Treatment Start
  Assessed via daily chest pain diary
Change in psychometric score at 3 months | 12 Weeks Post Treatment Start
  Assessed via SF-36 questionnaire and SCL-90 questionnaire.
Change in HRQOL scores at 3 months | 12 Weeks Post Treatment Start
  Assessed via health related quality of life (HRQOL) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Madanick, MD, Principal Investigator — UNC-Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States